



Study Number:

Patient Identification Number for this trial:

## **CONSENT FORM FOR RESEARCH STUDY**

**Title of Project:** "Success and survival of root canal treated tooth restored using ceramic onlays"

Name of Researcher: Noushad Rahim

## Please initial in the boxes to confirm

| • | | | inderstood the information sheet for the above study. |
|---|---|---|---|
| • | | | consider the information, ask nswered satisfactorily. |
| • | <ul> <li>I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected.</li> <li>I understand that relevant sections of any of my medical notes and data collected during the study may be looked at by responsible individuals from Guy's Hospital, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records.</li> </ul> | | |
| • | | | |
| • | I agree to take pa | rt in the above | research study. |
| Name of Patient | | Date | Signature |
| Name of Person Taking Consent | | Date | Signature |

When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes.